CLINICAL TRIAL: NCT03007251
Title: Immediate Effects of Eurythmy Therapy on Psychophysiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Jan Vagedes, Director and Head of the ARCIM Institute, ARCIM Institute Academic Research in Complementary and Integrative Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EYT_10
Record Dates: First submitted 2016-12-27; First posted 2017-01-02 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Eurythmy Therapy
MeSH Terms: interventions — Standing Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Eurythmy Therapy Movement "R" (Experimental): EYT exercise "R": Positioned between two steps and forearms parallel to the ground, the patient performs a rolling movement like wheels on a wagon. The movement is positioned below shoulder height and is initiated from the shoulder blade.
  Interventions: Other: Eurythmy Therapy Movement "R"
- Eurythmy Therapy Movement "L" (Experimental): EYT exercise "L": In a circular and flowing movement the patient leads his hands upwards in front of his body and down again laterally. During elevation of the arms, the patient performs a small hop onto the toes and into knock knees. Lowering his arms, he releases the legs and straightens up again.
  Interventions: Other: Eurythmy Therapy Movement "L"
- Eurythmy Therapy Movement "B" (Experimental): EYT exercise "B": The patient describes an embracing movement with both arms and the left leg while balancing on one foot. He then returns to the initial position and repeats the movement using the other leg.
  Interventions: Other: Eurythmy Therapy Movement "B"
- Normal movements during walking or standing (Active Comparator): Control exercise: Participants slowly walk across the room, their arms swinging in a natural way. This was designed to control for the most basic upright movement, shifting thermoregulation from resting conditions to exercise conditions, triggering non-thermal factors.
  Interventions: Other: Normal movements during walking or standing

INTERVENTIONS:
Other: Eurythmy Therapy Movement "R"
  Arms: Eurythmy Therapy Movement "R"
Other: Eurythmy Therapy Movement "L"
  Arms: Eurythmy Therapy Movement "L"
Other: Eurythmy Therapy Movement "B"
  Arms: Eurythmy Therapy Movement "B"
Other: Normal movements during walking or standing
  Arms: Normal movements during walking or standing

SUMMARY:
The purpose of this study is to investigate different effects of Eurythmy Therapy on psychological and physiological parameters of circulation and thermoregulation

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-55 Years old, signed informed consent available

Exclusion Criteria:

* Any known diseases of the cardiovascular system, allergic reactions to electrode patches in the past, coffee, alcohol or smoking less than 3 hours prior to the study, insufficient knowledge of the German language

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pulse Wave Velocity | 10 minutes after the movement exercises

IPD SHARING:
Plan to Share IPD: No